CLINICAL TRIAL: NCT02666677
Title: Invasive Instrumentation in Trauma Patients in the Shock Room: A Online-survey for Anaesthesia Departments in Germany
Brief Title: INVITE Study: Invasive Instrumentation in Trauma Patients in the Shock Room
Acronym: INVITE
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Köln (Other)
Collaborators: Universitätsklinikum Leipzig (Other); Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: INVITE
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Multiple Trauma
Keywords: polytrauma, emergency medicine
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is an online survey asking for invasive instrumention in trauma patients of an emergency department

DETAILED DESCRIPTION:
The INVITE study is an online survey for medical doctors asking for invasive instrumention (e.g., arterial line, entral venous line, etc.) in trauma patients of an emergency department

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple trauma
* treated in the emrgency department

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Traumatized patiennts in the emergency department
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2016-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
"Insertion of central venous catheter " survey | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Hinkelbein, MD, Principal Investigator — UK Köln
Locations (1):
- University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No